CLINICAL TRIAL: NCT06460272
Title: NOURISH HEARTS: Nutrition Outreach and Understanding: Research In Serving Hearts Through Healthy Eating And Tailored Support
Brief Title: Nutrition Outreach and Understanding: Research In Serving Hearts Through Healthy Eating And Tailored Support
Acronym: NOURISH HEARTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amanda Shallcross (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Amanda Shallcross, Director, Center for Research and Training, Department of Wellness and Preventative Medicine, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 24-472
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Type2diabetes; Metabolic Syndrome; Obesity
Keywords: Hypertension; Type2diabetes; Metabolic Syndrome; Obesity
MeSH Terms: conditions — Hypertension; Metabolic Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: This study is a human-centered three-arm design implementation trial to compare MTM only vs. MTM + SMA (weekly culinary and nutrition education and practice for 10 weeks) vs. a wait-list control group (MTM-Later). Meals will be provided at a frequency of 14 meals/week for 10 weeks. All intervention components will be designed and intended to be culturally congruent. Primary outcomes will be implementation (recruitment and retention rates) and feasibility (engagement and satisfaction).
  This study aims to distinguish an effective treatment (e.g., MTM only or MTM + SMAs) from a less effective or ineffective treatment. For this study, the investigators propose a three-arm (1:1:1) parallel-group randomized controlled trial (n = 75) powered to detect threshold levels of implementation and engagement. Intervention arms include, 1) MTM (only), 2) MTM +SMA, and a 3) Wait-list Control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and the study statistician will be masked to treatment condition when conducting initial data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medically Tailored Meals+ Shared Medical Appointments (MTMs + SMAs) (Experimental): Participants will receive 2 meals per day for 7 days a week for a duration of 10 weeks and SMA weekly for 10 weeks.
  Interventions: Other: Medically Tailored Meals
- Medically Tailored Meals (MTMs) (Active Comparator): Participants will receive 2 meals per day for 7 days a week for a duration of 10 weeks. Individuals randomized to MTMs will receive electronic educational materials from the MTM + SMA group after the completion of the post-intervention study assessment.
  Interventions: Other: Medically Tailored Meals
- Medically Tailored Meals - Later (MTM-Later) (Other): Participants will receive 2 meals per day for 7 days a week for a duration of 10 weeks and educational materials (e.g., relevant handouts from the SMA) after the completion of the post intervention study assessment. This group will act as our Waitlist Control group.
  Interventions: Other: Medically Tailored Meals

INTERVENTIONS:
Other: Medically Tailored Meals — Meals culturally tailored to provide essential nutrition

SUMMARY:
This study is a human-centered, three-arm, parallel-group, randomized control, implementation trial (n=75) to compare MTM (Medically Tailored Meals) only (14 meals delivered weekly for 10 weeks) vs. MTM + SMA (Shared Medical Appointments; once weekly sessions for 10 weeks) vs. a wait-list control group (MTM-Later) in patients with hypertension, type 2 diabetes, obesity, and/or metabolic syndrome. All intervention components will be culturally congruent (e.g., MTMs will include food that converges with culturally relevant diets and SMAs will be delivered by individuals with racial concordance to the target community). Primary outcomes will be implementation (recruitment and retention rates) and feasibility (engagement and satisfaction). Participants will be recruited from Cleveland Clinic's South Pointe Hospital in Warrensville Heights, a predominantly Black community with low socioeconomic status and high cardiovascular disease morbidity.

DETAILED DESCRIPTION:
Subjects will be randomized into one of the three arms within the study:

Medically Tailored Meals (MTMs):

Collaborative agreements are in place with Performance Kitchen to prepare 2 meals/day for 7 days/week for 10 weeks at a discount for all participants (n =75) for this trial. Meals will be prepared based on evidence-based nutritional recommendations for the Mediterranean diet and that align with 2021 American Heart Association Dietary Guidance. Individuals randomized to MTMs will receive electronic educational materials from the MTM + SMA group after the completion of the post-intervention study assessment.

Medically Tailored Meals + Shared Medical Appointments (MTMs + SMAs):

Identical MTMs that are provided in the MTM only group will also be provided in the MTM + SMA group. The SMA will be delivered weekly for 10 weeks and will be modeled after the investigator's pilot study. This includes practice with behavior change principles (i.e., selection of healthy food options). The provider, dietician, chef, and health coach will be members of the Black community to ensure racial concordance between educators and participants, a critical feature that improves communication, trust, and health outcomes in behavioral health interventions. The provider, dietician, and health coach are professionals currently employed within the Department of Wellness and Preventive Medicine. Fidelity will be ensured by using a session fidelity checklist that will be completed by each facilitator. To maximize retention, during consent via (telephone or in-person the study coordinator will establish rapport and set study expectations, including what SMAs entail and the time commitment for the session to minimize attrition. SMA visit reminder emails will be sent to participants through their EHR portal and/or via email.

Medically Tailored Meals - Later (MTM-Later):

The inclusion of a MTM-Later arm will provide a rigorous test of outcomes and is necessary given limited data about MTM implementation, engagement, and clinical outcomes in Black, underserved communities. MTM-Later participants will receive MTMs (same quantity and frequency) as the two other groups after the completion of the post-intervention study assessment. To avoid differential drop-out and incomplete assessments in the MTM-Later group, this group will be offered culinary tools at the start of the intervention to build trust and confidence that they will indeed receive the meals and educational materials at the end of the study assessment period. This group will act as the Waitlist Control group.

All groups will receive a set of surveys to be given at baseline and weeks 5 and 10 for exploratory outcomes. All groups will also have labs drawn at baseline and week 10 to measure secondary outcomes such as change in HbA1c.

4 focus groups will also be conducted (2 groups from each treatment arm) to understand barriers and facilitators to engaging in each of the active treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identification as Black or African American
2. Ability to speak and read English
3. Age ≥ 18 years old
4. Diagnosis of any of the following: a) Hypertension (>130/80), and ever treated for hypertension; b) Type 2 Diabetes Mellitus (HgbA1c ≥ 8%); c) Metabolic Syndrome; d) Obesity (BMI ≥ 30)
5. Access to a web-enabled device (phone, tablet, computer)
6. Received care at Cleveland Clinic South Pointe Hospital or Main Campus within the past 6 months

Exclusion Criteria:

1. Stage C and D heart failure
2. Advanced valvular heart disease
3. Advanced heart failure class D defined as heart failure symptoms impairing daily quality of life and/or resulting in recurrent hospitalizations (>1) per previous 12 months
4. Insulin requiring type II diabetes mellitus
5. Type I diabetes mellitus
6. Advanced chronic kidney disease (≥ Stage 4)
7. BMI > 45 kg/m2
8. Patients who are in another study or nutritional support program supplying meals
9. Patients who are receiving a medically prescribed diet with a specific nutritional profile
10. Receiving active cancer treatment, not including endocrine therapy
11. Inability to participate in the demands and requirements of the trial
12. Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Baseline through Week 10
  Recruitment is a measure of treatment implementation. Recruitment rate will be measured by # of participants enrolled in study/# passed eligibility screening.
Retention Rate | Baseline through Week 10
  Retention is a measure of treatment implementation. Retention rate will be measured by # of completed assessments at week 10/# randomized to treatment arm.
SMA Attendance | Baseline through Week 10
  Engagement will be assessed by Shared Medical Appointment (SMA) session attendance over the 10 week period.
MTMs Consumed | Baseline through Week 10
  Engagement will be assessed by proportion of Medically Tailored Meals (MTMs) consumed.
Satisfaction of the Intervention | Baseline through Week 10
  Satisfaction of MTM vs. MTM + SMA will be assessed using the Net Promoter Score (scale of 0 to 10; 9-10 being promoters, 7-8 being passives, and 0-6 being detractors)

SECONDARY OUTCOMES:
Eating Behavior | Baseline and Week 10
  Changes in eating behavior will be measured using the Mini-EAT (Eating Assessment Tool) and Fast Food/Restaurant Frequency Questionnaires.
Body Weight | Baseline and Week 10
  Body weight will be measured in pounds.
Waist/Hip Circumference | Baseline and Week 10
  Waist/Hip circumference will be expressed as a ratio.
Systolic and Diastolic Blood Pressure (mmHg) | Baseline and Week 10
  Systolic and diastolic blood pressure will be measured and expressed as mmHg.
Hemoglobin A1c (HbA1c, mmol/mol) | Baseline and Week 10
  Hemoglobin A1c will be evaluated through peripheral blood draw to assess diabetes control.
Trimethylamine N-oxide (TMAO, uM) | Baseline and Week 10
  Trimethylamine N-oxide will be evaluated through peripheral blood draw to assess cardiovascular disease risk.
Uric Acid (mg/dL) | Baseline and Week 10
  Uric Acid will be evaluated through peripheral blood draw to assess cardiovascular disease and diabetes risk.
Vitamin D 25 Hydroxy (ng/mL) | Baseline and Week 10
  Vitamin D 25 Hydroxy will be evaluated through peripheral blood draw to asses for Vitamin D deficiency.
High Sensitivity C-Reactive Protein (hsCRP, mg/dL) | Baseline and Week 10
  High Sensitivity C-Reactive Protein will be evaluated through peripheral blood draw to assess inflammation.

OTHER OUTCOMES:
Qualitative characterization of participants' lived experiences and engagement | Week 10
  4 focus groups (n=5 in each group, 2 groups from each treatment arm - MTM and MTM + SMA) will be conducted to understand barriers and facilitators to engaging in each of the active treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Shallcross, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Any factual data that is needed for independent verification of research results must be made freely and publicly available in an AHA-approved repository.
Supporting Information: Study Protocol
Time Frame: No later than the time of an associated publication or the end of the award period (and any no-cost extension), whichever come first.
Access Criteria: Individual participant data will become available at the conclusion of the study upon request by qualified individuals in the research community.

REFERENCES:
- [Background] Satia JA. Diet-related disparities: understanding the problem and accelerating solutions. J Am Diet Assoc. 2009 Apr;109(4):610-5. doi: 10.1016/j.jada.2008.12.019. No abstract available. PMID 19328255
- [Background] Eisenhauer E. In poor health: Supermarket redlining and urban nutrition. GeoJournal. 2001;53(2):125-133. doi:10.1023/A:1015772503007
- [Background] Black/African American Health-Office of Minority Health. Accessed October 24, 2023. https://minorityhealth.hhs.gov/blackafrican-american-health
- [Background] FastStats- Leading Causes of Death. Centers for Disease Control and Prevention. Published January 18, 2023. Accessed October 24, 2023. https://www.cdc.gov/nchs/fastats/leading-causes-of-death.htm
- [Background] Benjamins MR, Silva A, Saiyed NS, De Maio FG. Comparison of All-Cause Mortality Rates and Inequities Between Black and White Populations Across the 30 Most Populous US Cities. JAMA Netw Open. 2021 Jan 4;4(1):e2032086. doi: 10.1001/jamanetworkopen.2020.32086. PMID 33471116
- [Background] Belak L, Owens C, Smith M, Calloway E, Samnadda L, Egwuogu H, Schmidt S. The impact of medically tailored meals and nutrition therapy on biometric and dietary outcomes among food-insecure patients with congestive heart failure: a matched cohort study. BMC Nutr. 2022 Oct 3;8(1):108. doi: 10.1186/s40795-022-00602-y. PMID 36192812
- [Background] Berkowitz SA, Delahanty LM, Terranova J, Steiner B, Ruazol MP, Singh R, Shahid NN, Wexler DJ. Medically Tailored Meal Delivery for Diabetes Patients with Food Insecurity: a Randomized Cross-over Trial. J Gen Intern Med. 2019 Mar;34(3):396-404. doi: 10.1007/s11606-018-4716-z. Epub 2018 Nov 12. PMID 30421335
- [Background] Hager K, Cudhea FP, Wong JB, Berkowitz SA, Downer S, Lauren BN, Mozaffarian D. Association of National Expansion of Insurance Coverage of Medically Tailored Meals With Estimated Hospitalizations and Health Care Expenditures in the US. JAMA Netw Open. 2022 Oct 3;5(10):e2236898. doi: 10.1001/jamanetworkopen.2022.36898. PMID 36251292
- [Background] Berkowitz SA, Shahid NN, Terranova J, Steiner B, Ruazol MP, Singh R, Delahanty LM, Wexler DJ. "I was able to eat what I am supposed to eat"-- patient reflections on a medically-tailored meal intervention: a qualitative analysis. BMC Endocr Disord. 2020 Jan 20;20(1):10. doi: 10.1186/s12902-020-0491-z. PMID 31959176
- [Background] Winham DM. Culturally tailored foods and CVD prevention. Am J Lifestyle Med. 2009;3(1):64S-68S. doi: 10.1177/1559827609335552. PMID 20046905
- [Background] Bharmal N, Beidelschies M, Alejandro-Rodriguez M, Alejandro K, Guo N, Jones T, Bradley E. A nutrition and lifestyle-focused shared medical appointment in a resource-challenged community setting: a mixed-methods study. BMC Public Health. 2022 Mar 7;22(1):447. doi: 10.1186/s12889-022-12833-6. PMID 35255887
- [Background] Gardiner P, McGonigal L, Villa A, Kovell LC, Rohela P, Cauley A, Rinker D, Olendzki B. Our Whole Lives for Hypertension and Cardiac Risk Factors-Combining a Teaching Kitchen Group Visit With a Web-Based Platform: Feasibility Trial. JMIR Form Res. 2022 May 16;6(5):e29227. doi: 10.2196/29227. PMID 35576575
- [Background] Rohela P, Olendzki B, McGonigal LJ, Villa A, Gardiner P. A Teaching Kitchen Medical Groups Visit with an eHealth Platform for Hypertension and Cardiac Risk Factors: A Qualitative Feasibility Study. J Altern Complement Med. 2021 Nov;27(11):974-983. doi: 10.1089/acm.2021.0148. Epub 2021 Aug 5. PMID 34357790
- [Background] Lichtenstein AH, Appel LJ, Vadiveloo M, Hu FB, Kris-Etherton PM, Rebholz CM, Sacks FM, Thorndike AN, Van Horn L, Wylie-Rosett J. 2021 Dietary Guidance to Improve Cardiovascular Health: A Scientific Statement From the American Heart Association. Circulation. 2021 Dec 7;144(23):e472-e487. doi: 10.1161/CIR.0000000000001031. Epub 2021 Nov 2. PMID 34724806
- [Background] Moore C, Coates E, Watson A, de Heer R, McLeod A, Prudhomme A. "It's Important to Work with People that Look Like Me": Black Patients' Preferences for Patient-Provider Race Concordance. J Racial Ethn Health Disparities. 2023 Oct;10(5):2552-2564. doi: 10.1007/s40615-022-01435-y. Epub 2022 Nov 7. PMID 36344747
- [Background] Research methods: Is restricted randomisation necessary? Accessed June 1, 2021. https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1482349/
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Lara-Breitinger KM, Medina Inojosa JR, Li Z, Kunzova S, Lerman A, Kopecky SL, Lopez-Jimenez F. Validation of a Brief Dietary Questionnaire for Use in Clinical Practice: Mini-EAT (Eating Assessment Tool). J Am Heart Assoc. 2023 Jan 3;12(1):e025064. doi: 10.1161/JAHA.121.025064. Epub 2022 Dec 30. PMID 36583423
- [Background] ASA24 Dietary Assessment Tool- EGRP/DCCPS/NCI/NIH. Accessed October 23, 2023. https://epi.grants.cancer.gov/asa24/
- [Background] Medication History for Ambulatory-Surescripts. Accessed October 23, 2023. https://surescripts.com/what-we-do/medication-history-for-ambulatory
- [Background] Prescription Prices, Coupons & Pharmacy Information. GoodRx. Accessed October 23, 2023. https://www.goodrx.com/
- [Background] Woodward EN, Matthieu MM, Uchendu US, Rogal S, Kirchner JE. The health equity implementation framework: proposal and preliminary study of hepatitis C virus treatment. Implement Sci. 2019 Mar 12;14(1):26. doi: 10.1186/s13012-019-0861-y. PMID 30866982
- [Background] Gaglio B, Henton M, Barbeau A, Evans E, Hickam D, Newhouse R, Zickmund S. Methodological standards for qualitative and mixed methods patient centered outcomes research. BMJ. 2020 Dec 23;371:m4435. doi: 10.1136/bmj.m4435. PMID 33361103
- [Background] Diamond JJ. Development of a reliable and construct valid measure of nutritional literacy in adults. Nutr J. 2007 Feb 14;6:5. doi: 10.1186/1475-2891-6-5. PMID 17300716
- [Background] Cohen, S., Memelstein, R., Kamarck, T., & Hoberman, H. (1985). Measuring the functional components of social support. In I.G. Sarason & B. Sarason (Eds.), Social support: Theory, research and application (pp.73-94). The Hague: Martinus Nijhoff
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] Chen, G., Gully, S.M., & Eden, D. (2001). Validation of a new general self-efficacy scale. Organizational Research Methods, 4(1), 62-83
- [Background] Blumberg SJ, Bialostosky K, Hamilton WL, Briefel RR. The effectiveness of a short form of the Household Food Security Scale. Am J Public Health. 1999 Aug;89(8):1231-4. doi: 10.2105/ajph.89.8.1231. PMID 10432912
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Fernander AF, Duran RE, Saab PG, Llabre MM, Schneiderman N. Assessing the reliability and validity of the John Henry Active Coping Scale in an urban sample of African Americans and white Americans. Ethn Health. 2003 May;8(2):147-61. doi: 10.1080/13557850303563. PMID 14671768
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081